CLINICAL TRIAL: NCT06967376
Title: The Role of Adjuvant Cross Linking in the Management of Infective Keratitis - an OCT Based Assessment Study
Brief Title: The Role of Adjuvant Corneal Crosslinking in the Management of Infective Keratitis
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Research Institute of Ophthalmology, Egypt (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RIO Egypt (approval number 109
Record Dates: First submitted 2024-11-02; First posted 2025-05-13 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2024-11

CONDITIONS: Infective Keratitis
MeSH Terms: interventions — Anti-Infective Agents

STUDY DESIGN:
Intervention Model Description: Methods
  Study Design:
  A prospective, single centre, randomised controlled study of forty eyes of forty patients was conducted. The study was approved by local institutional review board (Approval number 109) and adhered to the Declaration of Helsinki. All patients provided informed consent before enrolling and participating in the study.
  Selection:
  All patients presenting with infective keratitis were explained about the study and informed consent was sought (CONSORT Diagram). Fifty-three patients were screened against the exclusion criteria and 13 were excluded. The remaining total of 40 patients were allocated equally to two groups (A and B) by process of simple randomisation. Group A patients were to be offered standard targeted anti-microbial therapy whilst group B were offered CXL in addition to the standard targeted anti-microbial therapy.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Arm that take medical treatment only for infective keratitis (Active Comparator): On presentation, all pre-existing treatment was stopped for 48 hours and corneal scrapes for direct smears and cultures using blood agar, chocolate agar, thioglycolate broth and sabouraud dextrose agar were done. Initial antimicrobial therapy for both groups consisted of fortified vancomycin eye drops 50 mg/ml, fortified ceftazidime eye drops 50 mg/ml hourly, and the antifungal agent itraconazole 100 mg orally twice per day. This regimen was subject to change according to microbiology culture sensitivities and/or results.
  Interventions: Drug: Topical Antimicrobial/Antifungal Medications
- Arm of patients take cross linking as an adjuvant treatment to medical treatment (Active Comparator): Patients allocated to the PACK-CXL group were assessed and treated by PACK-CXL within 2 days of treatment initiation. Topical anaesthesia was achieved using 0.4% benoxinate hydrochloride drops. Epithelium was removed up to 9 mm diameter. Corneal thickness of the area to be treated was measured (without epithelium) aiming for a starting thickness of no less than 350μm. Corneas thicker than 500μm were dehydrated to reduce thickness by using 70% Glycerol drops applied topically at intervals of 2-3 seconds for a total of five minutes. A schematic representation of PACK-CXL protocol is provided in Figure 1. Iso-osmolar riboflavin drops were instilled topically on the cornea at regular intervals of 2 minutes for a total period of 30 minutes. Thickness was also re-measured every 5 min to ensure that it remained below 500µm during instillation of riboflavin. The cornea was illuminated using a UVX, UV-A 365 nm with an irradiance of 3 mW/cm2 for 30 minutes and a total dose of 5.4 J/cm2 during
  Interventions: Procedure: Corneal Collagen Cross-Linking Solutions

INTERVENTIONS:
Procedure: Corneal Collagen Cross-Linking Solutions — Topical anaesthesia was achieved using 0.4% benoxinate hydrochloride drops. Epithelium was removed up to 9 mm diameter. Corneal thickness of the area to be treated was measured (without epithelium) aiming for a starting thickness of no less than 350μm. Corneas thicker than 500μm were dehydrated to reduce thickness by using 70% Glycerol drops applied topically at intervals of 2-3 seconds for a total of five minutes. A schematic representation of PACK-CXL protocol is provided in Figure 1. Iso-osmolar riboflavin drops were instilled topically on the cornea at regular intervals of 2 minutes for a total period of 30 minutes. Thickness was also re-measured every 5 min to ensure that it remained below 500µm during instillation of riboflavin. The cornea was illuminated using a UVX, UV-A 365 nm with an irradiance of 3 mW/cm2 for 30 minutes and a total dose of 5.4 J/cm2 during which riboflavin was instilled every 2 min and corneal pachymetry performed every 5 min. PACK-CXL was performed in a 9
  Arms: Arm of patients take cross linking as an adjuvant treatment to medical treatment
Drug: Topical Antimicrobial/Antifungal Medications — Initial antimicrobial therapy for both groups consisted of fortified vancomycin eye drops 50 mg/ml, fortified ceftazidime eye drops 50 mg/ml hourly, and the antifungal agent itraconazole 100 mg orally twice per day. This regimen was subject to change according to microbiology culture sensitivities and/or results.
  Arms: Arm that take medical treatment only for infective keratitis

SUMMARY:
This was a prospective, single centre, randomised controlled study to evaluate the clinical effectiveness of corneal collagen crosslinking as an adjuvant to antimicrobial therapy.

DETAILED DESCRIPTION:
This randomised controlled study of forty eyes of forty patients was conducted to assess the impact of corneal collagen crosslinking in addition to antimicrobial therapy.

All forty patients presenting with infective keratitis of various aetiologies (bacterial, fungal, acanthamoeba) were screened and then randomly allocated equally to two groups (A and B). Group A patients were to be offered standard targeted anti-microbial therapy whilst group B were offered CXL in addition to the standard targeted anti-microbial therapy.

Patients were evaluated clinically for visual acuity; infection parameters and dimensions were measured on slit lamp and optical coherence tomography. Evaluations were noted at the baseline visit and subsequently on days 7, 14, and day 30 of treatment

ELIGIBILITY:
Inclusion Criteria:

• Patients presenting with infectious keratitis

Exclusion Criteria:

* Infective keratitis < 1mm from limbus
* Corneal thickness < 350μm
* Previous herpetic eye disease
* Expectant and nursing women

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-05-21 (Actual); Primary Completion 2021-11-11 (Actual); Study Completion 2022-02-03 (Actual)

PRIMARY OUTCOMES:
clinical response | At presentation; and then on day 7, day 14 and day 30 of commencing treatment
  Ulcer dimensions will be studied on slit lamp and AS-OCT.

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Research Institute of Ophthalmology, Giza, Giza Governorate
  - Research Institute of Ophthalmology, Giza

IPD SHARING:
Plan to Share IPD: No